CLINICAL TRIAL: NCT02194439
Title: Bridging Pediatric and Adult Biomarkers in Graft-Versus-Host Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sophie Paczesny, Professor of Pediatrics and Immunology, Indiana University
Other Study IDs: 1405976232; 1R01HD074587-01 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-18 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Graft-Versus-Host Disease
Keywords: Acute Graft Versus Host Disease; Affect; Anti-inflammatory; Anti-inflammatory Agents; Antigen-Presenting Cells; Alloantigen; Allogeneic; Allograft rejection; Allograft Tolerance; Antigens; Autoimmunity; Biomarkers; Biospecimen Repository; BMT; Bone Marrow Transplantation; Cell Transplantation; Cells; Clonal Expansion; Complex; Cytokine; Data; Development; Environment; Failure (biologic function); Genomics; Graft-vs-Host Disease; Graft-vs-Leukemia; GVHD; GVL; Hematopoietic; Hematopoietic Stem Cell Transplantation; HCT; HSCT; IL-33 Receptor; Immune Reconstitution; Immune Response; Inflammatory; Modeling; Novel; Novel therapeutics; Outcome; Pathway interactions; Peptides; Prevent; Process; Production; Proteomics; Regulatory T-Lymphocyte; Response; Role; Signal; ST2; Transduction; T-cell response; T-cell Activation; T-Lymphocytes; Tissues
MeSH Terms: conditions — Graft vs Host Disease; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Plasma, Peripheral Blood Mononuclear Cells (PBMC), Saliva, Bronchoalveolar lavage (BAL)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hematopoietic stem cell transplant: procedure

SUMMARY:
This study is designed to collect longitudinal biological samples from patients after hematopoietic cell transplantation (HCT) cared for at multiple bone marrow transplant centers to validate biomarkers of both acute and chronic GVHD as well as for use in future unspecified research. The centers include Dana-Farber Cancer Institute and Boston's Children's Hospital, Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Fred Hutchinson Cancer Research Center, Texas Children's Hospital, Children's National Medical Center, and Indiana University Simon Cancer Center.

DETAILED DESCRIPTION:
After informed consent is signed, this study will involve 1) collection of basic HCT data and clinical data available in the medical record and 2) providing blood (and saliva in occasional cases) samples for processing, storage, DNA extraction, and analysis (including a seven biomarker protein panel as well as future unspecified research purposes).

Pediatric and adult patients will be included (all adult patients will be from the Fred Hutchinson Cancer Research Center, the Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, and the Indiana University Simon Cancer Center).

Primary Objective:

1. To confirm that ST2 alone or the seven-biomarker panel measured at initiation of GVHD therapy predict a) D180 post-therapy non-relapse mortality; b) D28 post-therapy non-response, and c) GVHD grade 1-4 onset D180 post-therapy non-relapse mortality.

Secondary Objective:

1. To demonstrate that ST2 alone or the seven-biomarker panel measured at day 14 or day 21 post-HCT (or a combination of these time points) predicts D180 post-HCT non-relapse mortality.
2. To demonstrate that ST2 alone or the seven-biomarker panel measured at initiation of GVHD symptoms/therapy diagnose acute GVHD as compared to other complications presenting with similar symptoms (drug rash, CMV, Clostridium enteritis).
3. To demonstrate that ST2 alone or the seven-biomarker panel measured at initiation of GVHD symptoms/therapy diagnose the severity of acute GVHD at onset and maximum.
4. To develop a repository of biospecimens linked to clinical data for future unspecified research.

ELIGIBILITY:
Inclusion Criteria: - All patients receiving an allogeneic hematopoietic stem cell transplant, cord blood transplant, bone marrow transplant, T cell depleted marrow, donor lymphocyte infusion (DLI), or donor cellular infusion (DCI) can be included.

Exclusion Criteria: - patients not receiving an allogeneic hematopoietic stem cell transplant, cord blood transplant, bone marrow transplant, T cell depleted marrow, donor lymphocyte infusion (DLI), or donor cellular infusion (DCI) will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients receiving an allogeneic hematopoietic stem cell transplant, cord blood transplant, bone marrow transplant, T cell depleted marrow, donor lymphocyte infusion (DLI), or donor cellular infusion (DCI) from Dana-Farber Cancer Institute and Boston Children's Hospital, Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Fred Hutchinson Cancer Research Center, Texas Children's Hospital, Children's National Medical Center, and Indiana University Simon Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Paczesny, MD, PhD, Study Chair — Indiana University
Locations (1):
- Indiana Unversity Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Rowan CM, Pike F, Cooke KR, Krance R, Carpenter PA, Duncan C, Jacobsohn DA, Bollard CM, Cruz CRY, Malatpure A, Farag SS, Renbarger J, Liu H, Bakoyannis G, Hanash S, Paczesny S. Assessment of ST2 for risk of death following graft-versus-host disease in pediatric and adult age groups. Blood. 2020 Apr 23;135(17):1428-1437. doi: 10.1182/blood.2019002334. PMID 31972009

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplant: 4 plasma biomarkers were assessed pre-HCT and at days +7, +14 and +21 post-HCT.
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplant
Started | 415
Completed | 415
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who performed biomarker collection.
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 415
Age, Customized [Count of Participants; unit: Participants]
  Age <10 | 170
  Age >10 | 245
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55
  Not Hispanic or Latino | 351
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 51
  White | 293
  More than one race | 40
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 415

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non Relapse Mortality (NRM) by Age and ST2 at 12 Months Post-HCT
Description: To measure stimulation-2 (ST2) pre-HCT by number of participants at 12 months post-HCT for non-relapse mortality according to ST2 values and age less than or equal to 10 and greater than 10 using landmark analyses.
Time Frame: 1 year
Population: Participants who had all four biomarkers and four timepoints.
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 415
participants
  Age <10 high Pre-HCT ST2 >26 | 55
  Age <10 low pre-HCT ST2 <26 | 115
  Age >10 high Pre-HCT ST2 >26 | 125
  Age >10 low Pre-HCT ST2 <26 | 120

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Hematopoietic Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 0/415
Serious Adverse Events (participants affected / at risk) | 0/415
Other Adverse Events (participants affected / at risk) | 0/415

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT02194439/SAP_000.pdf
  • Study Protocol (2015-06-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02194439/Prot_001.pdf